CLINICAL TRIAL: NCT02833662
Title: Evolution of the Severity of Obstructive Sleep Apnea and Consequences on Cardiac Rhythm Abnormalities After Surgery Under General Anesthesia
Brief Title: Evaluation of Sleep Apnea and Cardiac Rhythm Abnormalities After Surgery Under General Anesthesia
Acronym: Etude3A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 38RC15.080
Record Dates: First submitted 2015-06-03; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea; Arrhythmia
Keywords: Hypoxia; Perioperative outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Arrhythmias, Cardiac; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients suspected to present a Sleep Apnea Syndrom (Other): Record nocturnal respiratory and cardiac parameters before and after surgery :
  Severity of sleep respiratory disorders and relationship with cardiac rhythm abnormalities will be assessed in patients suspected to present Sleep Apnea, before and after surgery under general anesthesia.
  Interventions: Other: Measure of ODI and heart rhythm

INTERVENTIONS:
Other: Measure of ODI and heart rhythm — Record nocturnal respiratory and cardiac parameters before and after surgery.

SUMMARY:
Higher risk of cardiac and respiratory post-operative events is observed in patients with unrecognised Obstructive Sleep Apnea (OSA). The efficiency of a simple method of OSA screening by analysing ventilation with measurement of nose pressure and nocturnal hypoxemia (oxygen desaturation index) will be assessed. These sleep respiratory analyses will be compared with the research of arrhythmia, in order to show if they are linked to the hypoxemia events.

Aggravation of nocturnal respiratory disorder and higher incidence of cardiac and respiratory postoperative complications will be assessed in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* orthopaedic, urologic, vascular, digestive surgery
* under general anaesthesia or sedation
* age > 45 years old
* STOP-BANG score>3

Exclusion Criteria:

* Head and neck surgery, planned prolonged mechanical ventilation after surgery (>24h)
* Severe COPD
* Post-operative ICU planned
* Diagnosed OSA or other sleep disorder breathing

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in heart rhythm troubles linked to hypoxemia events | Before surgery and at first and third night after surgery
  Heart rhythm troubles will be assessed 3 times:
  * First time = baseline assessment, during one night before surgery
  * second assessment will occur during the first night after surgery
  * last assessment will take place during the third night after surgery

SECONDARY OUTCOMES:
Change from baseline in severity of OSA defined by the oxygen saturation index | Before surgery and at first and third night after surgery
  OSA will be assessed 3 times:
  * First time = baseline assessment, during one night before surgery
  * second assessment will occur during the first night after surgery
  * last assessment will take place during the third night after surgery oxygen saturation index > 10 mandatory for the study oxygen saturation index > 40 : result qualified severe
Aggravation of cardiac events linked to hypoxemia | After surgery from night 1 to night 15 maximum
Change from baseline OSA prevalence and cardiorespiratory complications after surgery | Before surgery and at first and third night after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, Md,PhD, Principal Investigator — University Hospital, Grenoble

REFERENCES:
- [Background] Chung F, Liao P, Yegneswaran B, Shapiro CM, Kang W. Postoperative changes in sleep-disordered breathing and sleep architecture in patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):287-98. doi: 10.1097/ALN.0000000000000040. PMID 24158049
- [Background] Kaw R, Chung F, Pasupuleti V, Mehta J, Gay PC, Hernandez AV. Meta-analysis of the association between obstructive sleep apnoea and postoperative outcome. Br J Anaesth. 2012 Dec;109(6):897-906. doi: 10.1093/bja/aes308. Epub 2012 Sep 6. PMID 22956642
- [Background] Vizzardi E, Sciatti E, Bonadei I, D'Aloia A, Curnis A, Metra M. Obstructive sleep apnoea-hypopnoea and arrhythmias: new updates. J Cardiovasc Med (Hagerstown). 2017 Jul;18(7):490-500. doi: 10.2459/JCM.0000000000000043. PMID 25000252
- [Background] Kilicaslan F, Tokatli A, Ozdag F, Uzun M, Uz O, Isilak Z, Yiginer O, Yalcin M, Guney MS, Cebeci BS. Tp-e interval, Tp-e/QT ratio, and Tp-e/QTc ratio are prolonged in patients with moderate and severe obstructive sleep apnea. Pacing Clin Electrophysiol. 2012 Aug;35(8):966-72. doi: 10.1111/j.1540-8159.2012.03439.x. Epub 2012 Jun 5. PMID 22671991
- [Background] Chung F, Liao P, Elsaid H, Shapiro CM, Kang W. Factors associated with postoperative exacerbation of sleep-disordered breathing. Anesthesiology. 2014 Feb;120(2):299-311. doi: 10.1097/ALN.0000000000000041. PMID 24158050
- [Background] Singh M, Liao P, Kobah S, Wijeysundera DN, Shapiro C, Chung F. Proportion of surgical patients with undiagnosed obstructive sleep apnoea. Br J Anaesth. 2013 Apr;110(4):629-36. doi: 10.1093/bja/aes465. Epub 2012 Dec 19. PMID 23257990
- [Background] Rennotte MT, Baele P, Aubert G, Rodenstein DO. Nasal continuous positive airway pressure in the perioperative management of patients with obstructive sleep apnea submitted to surgery. Chest. 1995 Feb;107(2):367-74. doi: 10.1378/chest.107.2.367. PMID 7842763
- [Background] Latina JM, Estes NA 3rd, Garlitski AC. The Relationship between Obstructive Sleep Apnea and Atrial Fibrillation: A Complex Interplay. Pulm Med. 2013;2013:621736. doi: 10.1155/2013/621736. Epub 2013 Feb 26. PMID 23533751
- [Background] Gupta S, Cepeda-Valery B, Romero-Corral A, Shamsuzzaman A, Somers VK, Pressman GS. Association between QRS duration and obstructive sleep apnea. J Clin Sleep Med. 2012 Dec 15;8(6):649-54. doi: 10.5664/jcsm.2256. PMID 23243398
- [Background] Filgueiras-Rama D, Arias MA, Iniesta A, Armada E, Merino JL, Peinado R, Lopez-Sendon JL. Atrial arrhythmias in obstructive sleep apnea: underlying mechanisms and implications in the clinical setting. Pulm Med. 2013;2013:426758. doi: 10.1155/2013/426758. Epub 2013 Apr 3. PMID 23691306
- [Background] Rossi VA, Stradling JR, Kohler M. Effects of obstructive sleep apnoea on heart rhythm. Eur Respir J. 2013 Jun;41(6):1439-51. doi: 10.1183/09031936.00128412. Epub 2012 Dec 20. PMID 23258782
- [Background] Gami AS, Olson EJ, Shen WK, Wright RS, Ballman KV, Hodge DO, Herges RM, Howard DE, Somers VK. Obstructive sleep apnea and the risk of sudden cardiac death: a longitudinal study of 10,701 adults. J Am Coll Cardiol. 2013 Aug 13;62(7):610-6. doi: 10.1016/j.jacc.2013.04.080. Epub 2013 Jun 13. PMID 23770166
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Background] Chouchou F, Poupard L, Philippe C, Court-Fortune I, Barthelemy JC, Roche F. Thoracic impedance, in association with oximetry, in a multi-modal ECG Holter system is useful for screening sleep disordered breathing. Int J Cardiol. 2013 Feb 10;163(1):100-2. doi: 10.1016/j.ijcard.2012.06.082. Epub 2012 Jul 16. No abstract available. PMID 22805548
- [Background] Poupard L, Mathieu M, Goldman M, Chouchou F, Roche F. Multi-modal ECG Holter system for sleep-disordered breathing screening: a validation study. Sleep Breath. 2012 Sep;16(3):685-93. doi: 10.1007/s11325-011-0558-1. Epub 2011 Jul 26. PMID 21789729
- [Background] Baguet JP, Levy P, Barone-Rochette G, Tamisier R, Pierre H, Peeters M, Mallion JM, Pepin JL. Masked hypertension in obstructive sleep apnea syndrome. J Hypertens. 2008 May;26(5):885-92. doi: 10.1097/HJH.0b013e3282f55049. PMID 18398330
- [Background] Pepin JL, Defaye P, Vincent E, Christophle-Boulard S, Tamisier R, Levy P. Sleep apnea diagnosis using an ECG Holter device including a nasal pressure (NP) recording: validation of visual and automatic analysis of nasal pressure versus full polysomnography. Sleep Med. 2009 Jun;10(6):651-6. doi: 10.1016/j.sleep.2008.07.002. Epub 2008 Nov 22. PMID 19028140
- [Background] Tamisier R, Gilmartin GS, Launois SH, Pepin JL, Nespoulet H, Thomas R, Levy P, Weiss JW. A new model of chronic intermittent hypoxia in humans: effect on ventilation, sleep, and blood pressure. J Appl Physiol (1985). 2009 Jul;107(1):17-24. doi: 10.1152/japplphysiol.91165.2008. Epub 2009 Feb 19. PMID 19228987
- [Background] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795
- [Background] Tamisier R, Pepin JL, Remy J, Baguet JP, Taylor JA, Weiss JW, Levy P. 14 nights of intermittent hypoxia elevate daytime blood pressure and sympathetic activity in healthy humans. Eur Respir J. 2011 Jan;37(1):119-28. doi: 10.1183/09031936.00204209. Epub 2010 Jun 4. PMID 20525723
- [Background] Roche F, Pepin JL, Achour-Crawford E, Tamisier R, Pichot V, Celle S, Maudoux D, Chouchou F, Ntougou-Assoumou HG, Levy P, Barthelemy JC; PROOF Study Group. At 68 years, unrecognised sleep apnoea is associated with elevated ambulatory blood pressure. Eur Respir J. 2012 Sep;40(3):649-56. doi: 10.1183/09031936.00162710. Epub 2012 Apr 20. PMID 22523363
- [Background] Cereda CW, Tamisier R, Manconi M, Andreotti J, Frangi J, Pifferini V, Bassetti CL. Endothelial dysfunction and arterial stiffness in ischemic stroke: the role of sleep-disordered breathing. Stroke. 2013 Apr;44(4):1175-8. doi: 10.1161/STROKEAHA.111.000112. Epub 2013 Mar 7. PMID 23471270
- [Background] Gasa M, Tamisier R, Launois SH, Sapene M, Martin F, Stach B, Grillet Y, Levy P, Pepin JL; Scientific Council of the Sleep Registry of the French Federation of Pneumology-FFP. Residual sleepiness in sleep apnea patients treated by continuous positive airway pressure. J Sleep Res. 2013 Aug;22(4):389-97. doi: 10.1111/jsr.12039. Epub 2013 Feb 15. PMID 23409736
- [Background] Maziere S, Pepin JL, Siyanko N, Bioteau C, Launois S, Tamisier R, Arnol N, Levy P, Couturier P, Bosson JL, Gavazzi G. Usefulness of oximetry for sleep apnea screening in frail hospitalized elderly. J Am Med Dir Assoc. 2014 Jun;15(6):447.e9-14. doi: 10.1016/j.jamda.2014.03.011. Epub 2014 Apr 24. PMID 24768555
- [Background] Minville C, Hilleret MN, Tamisier R, Aron-Wisnewsky J, Clement K, Trocme C, Borel JC, Levy P, Zarski JP, Pepin JL. Nonalcoholic fatty liver disease, nocturnal hypoxia, and endothelial function in patients with sleep apnea. Chest. 2014 Mar 1;145(3):525-533. doi: 10.1378/chest.13-0938. PMID 24264333
- [Derived] Seguin L, Mendelson M, Doutreleau S, Clin R, Destors M, Albaladejo P, Pepin JL, Payen JF, Tamisier R. Temporal link between cardiac arrhythmias and postoperative episodes of hypoxemia during nocturnal sleep in patients with obstructive sleep apnea syndrome. Sleep Med. 2024 Dec;124:260-267. doi: 10.1016/j.sleep.2024.09.014. Epub 2024 Sep 12. PMID 39332270
- [Derived] Seguin L, Tamisier R, Deletombe B, Lopez M, Pepin JL, Payen JF. Preoperative Screening for Obstructive Sleep Apnea Using Alternative Scoring Models of the Sleep Tiredness Observed Pressure-Body Mass Index Age Neck Circumference Gender Questionnaire: An External Validation. Anesth Analg. 2020 Oct;131(4):1025-1031. doi: 10.1213/ANE.0000000000004909. PMID 32925319